CLINICAL TRIAL: NCT01132651
Title: Novel Use of a Cooling Pillow for Treatment of Severe Hand and Neck Atopic Dermatitis
Brief Title: Cooling Pillow for Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dennis West, Professor in Dermatology and Pediatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 28933
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: eczema; itch; pruritus; head; neck
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chillow cooling pillow (Experimental): This group of subjects will follow their current eczema regimen with the addition of using the cooling pillow at night to sleep on.
  Interventions: Other: Chillow cooling pillow
- Standard of care (regular pillow at night) (Placebo Comparator): This group of subjects will serve as the control group following a their current eczema care regimen, including sleeping on their normal pillow.
  Interventions: Other: Current standard eczema treatment and standard pillow at night

INTERVENTIONS:
Other: Current standard eczema treatment and standard pillow at night — Subjects will continue with their current eczema care and use their normal pillow at night.
  Arms: Standard of care (regular pillow at night)
Other: Chillow cooling pillow — Subjects will use the cooling pillow to sleep on in addition to their current eczema treatment for 2 weeks.
  Arms: Chillow cooling pillow

SUMMARY:
The purpose of this study is to see if using a cooling pillow at night will help sleep quality in people with atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD by dermatologist
* AD located on the head and neck
* Investigator Global Assessment (IGA)score >3 at time of enrollment
* Able to read, write, and understand study materials
* Age 18 or older

Exclusion Criteria:

* Concurrent non-AD skin disease on the head and neck
* Active skin infection on the head and neck, or conditions that may interfere with evaluation of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis West, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chillow (Cooling Pillow): This group of subjects followed their current eczema regimen with the addition of sleeping on the cooling pillow at night.
- Control (Normal Pillow): This group of subjects served as the control group. They followed their current eczema regimen and slept on their normal pillow at night.
Period: Overall Study
Arm/Group | Chillow (Cooling Pillow) | Control (Normal Pillow)
Started | 4 | 5
Completed | 3 | 4
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chillow (Cooling Pillow) | Control (Normal Pillow) | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.3) | 34 (13.5) | 34.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep Quality as Measured by a Change in Pittsburgh Sleep Quality Index (PSQI) Survey Score
Description: The PSQI is a clinical survey used to measure sleep quality. Seven components related to sleep quality are scored: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Each component is scored on a scale of 0 to 3. A score of 0 is associated with better sleep quality and a score of 3 is associated with worse sleep quality. The seven component scores are summed to achieve a total PSQI score. The total PSQI score has a range of 0-21. A score of 0 is associated with better sleep quality and a score of 21 is associated with worse sleep quality.
  Buysse,D.J., Reynolds,C.F., Monk,T.H., Berman,S.R., & Kupfer,D.J. (1989). The Pittsburgh Sleep Quality Index (PSQI): A new instrument for psychiatric research and practice. Psychiatry Research, 28(2), 193-213.
Time Frame: Baseline and at 2 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Chillow (Cooling Pillow) | Control (Normal Pillow)
Number analyzed (Participants) | 3 | 4
units on a scale | -1 [-2 to 0] | -2 [-3 to 2]

2. Secondary Outcome: Change in Severity of Atopic Dermatitis (AD) as Measured by a Change in Investigator Global Assessment (IGA) Score
Description: The IGA score is an assessment of AD severity. It is an assessment of the patient's disease state at the time of examination and does not attempt a comparison with any of the patient's previous disease states. Possible scores range from 0 to 5. A score of 0 is associated with no evidence of AD and a score of 5 is associated with severe AD.
Time Frame: Baseline and at 2 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Chillow (Cooling Pillow) | Control (Normal Pillow)
Number analyzed (Participants) | 3 | 4
units on a scale | -1 [-1 to -1] | -1 [-2 to 0]

ADVERSE EVENTS:
Arm/Group | Chillow (Cooling Pillow) | Control (Normal Pillow)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes